CLINICAL TRIAL: NCT05722119
Title: Clinical Impact of the BioFire gastroIntestinal Panel for the Management of Diarrhea in Kidney Transplant Patients
Brief Title: GastroIntestinal Panel in Kidney Transplant Patients
Acronym: GIPIK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP211588
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Kidney Transplant; Complications; Diarrhoea;Acute; Diarrhea Infectious
MeSH Terms: conditions — Dysentery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiplex test (Experimental): Multiplex Polymerase Chain Reaction (PCR) assay on stool samples, within 2 hours, in patients with acute diarrhea
  Interventions: Diagnostic Test: FilmArray GI
- Standard of care tests (No Intervention): Coproculture with direct examination and Clostridium difficile and A-B toxins search, parasitological examination of the stool and search for enteric viruses (rotavirus, adenovirus, norovirus, astrovirus) in patients with acute diarrhea
- Control group without diarrhea (Experimental): Multiplex Polymerase Chain Reaction (PCR) assay on stool samples in asymptomatic patients
  Interventions: Diagnostic Test: FilmArray GI

INTERVENTIONS:
Diagnostic Test: FilmArray GI — Rapid multiplex Polymerase Chain Reaction (PCR) assay for digestive infectious agents in stool sample in the baseline diagnostic tests panel
  Other Names: Multiplex Polymerase Chain Reaction (PCR) assay
  Arms: Control group without diarrhea; Multiplex test

SUMMARY:
This project focuses on the evaluation of the impact of the rapid mutltiplex test on changes in anti-infectious treatments in kidney transplant patients with diarrhea. A higher number of infectious agents detected on the same day of sampling could improve the etiological diagnosis of diarrhea in kidney transplant patients and optimize therapeutic management.

A prospective study will be conducted to evaluate the impact of a rapid multiplex test with a wide panel of bacteria, viruses and parasites on the clinical management of kidney transplant patients with acute diarrhea. This impact will be evaluated using a control group of kidney transplant patients with acute diarrhea whose infectious diagnosis will be performed by standard methods. The main objective is to determine the impact of the rapid multiplex test on changes in anti-infectious treatments (initiation, change of molecule, total duration of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent
* Patient who received a kidney transplant at least 3 months ago
* Acute diarrhea (at least 3 unformed or liquid stools per day for at least 3 consecutive days or 3 per day and / or weight loss ≥2 kg and / or mucoid and / or bloody stool) or absence of diarrhea for at least a month (asymptomatic non randomized control group)
* Affiliation to social security in accordance with the recommendations of the French law

Exclusion Criteria:

* Patients who received an identical HLA transplant from a related donor
* Patients without health insurance
* Patients under guardianship or curatorship
* Pregnant (or breastfeeding) patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Difference in the proportion of patients with anti-infectious treatment change | 1 week
  Difference in the proportion of patients with an adapation of anti-infectious treatment between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Difference in the time to anti-infectious treatment change | 1 week
  Difference in the time to an adaptation of anti-infectious treatment between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)

SECONDARY OUTCOMES:
Difference in the proportion of patients with an adaptation of immunosuppressive therapy | 30 days
  Difference in the proportion of patients with an adaptation of immunosuppressive therapy between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Difference in the time to adaptation of immunosuppressive therapy | 30 days
  Difference in the time to adaptation of immunosuppressive therapy between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Proportion of patients with additional tests for the etiological diagnosis of diarrhea | 30 days
  Difference in the proportion of patients with additional tests for the etiological diagnosis of diarrhea between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Number of additional tests for the etiological diagnosis of diarrhea | 30 days
  Difference in the number additional tests for the etiological diagnosis of diarrhea between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Time to digestive endoscopy | 30 days
  Difference in the time to digestive endoscopy between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Duration of diarrhea | 30 days
  Difference in the duration of diarrhea between the 2 randomized groups (rapid multiplex test group versus standard tests in patients with acute diarrhea)
Proportion of patients with asymptomatic carriage of infectious agents | Day 1
  Proportion of patients with asymptomatic carriage of infectious agents in the asymptomatic control group
Quantitative polymerase chain reaction (PCR) by multiplex PCR for infectious agents | Day 1
  Quantitative polymerase chain reaction (PCR) by multiplex PCR for infectious agents on a stool sample at baseline
Alpha-diversity | Day 1
  Microbiota alpha-diversity on a stool sample at baseline
Beta-diversity | Day 1
  Microbiota beta-diversity on a stool sample at baseline

IPD SHARING:
Plan to Share IPD: Undecided